CLINICAL TRIAL: NCT06341231
Title: Personalized Anticoagulant Therapy for Pulmonary Thromboembolism in Specific Populations With Older Age, Renal Insufficiency or Co-existing Malignancy
Brief Title: Personalized Anticoagulant Therapy for Pulmonary Thromboembolism
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 202400248
Record Dates: First submitted 2024-03-12; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Thromboembolisms; Anticoagulants; Increased
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Elderly patients with pulmonary thromboembolism
- Pulmonary thromboembolism patients with renal insufficiency
- Pulmonary thromboembolism patients with co-existing malignancy

SUMMARY:
The goal of this prospective observational study is to explore the influencing factors of the efficacy and safety of anticoagulant therapy for pulmonary thromboembolism in special populations with older age, renal insufficiency or co-existing malignancy, and establish a predictive model to guide clinical practice. The main questions it aims to answer are:

* To analyze the influencing factors of the efficacy and safety of anticoagulant therapy for specific populations with pulmonary thromboembolism (PTE) in the real world (such as the elderly, those with impaired kidney function, and individuals with malignant tumors).
* Whether we can use machine-learning models to predict bleeding events and VTE recurrence in special populations following anticoagulant therapy in the real world? Participants will receive diagnostic and therapeutic measures for pulmonary thromboembolism in accordance with clinical guidelines, including anticoagulant therapy. Some patients need to have peripheral blood samples collected at the time of enrollment and 3 months after anticoagulant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Adult patients with objectively diagnosed pulmonary thromboembolism (PTE) (with or without concomitant deep vein thrombosis);
3. Specific populations meeting any of the following criteria: elderly patients (≥75 years old); patients with impaired kidney function (creatinine clearance estimated by the Cockcroft-Gault formula, CrCl < 60ml/min); patients with active malignancies (under treatment or with unrecovered malignancies);
4. Patients who have not started anticoagulant therapy before enrollment and are planned for anticoagulant treatment after evaluation by the attending physician;
5. Ecpected life expectancy longer than 3 months.
6. Patients who understand and agree to participate in this study, sign the informed consent form, and adhere to regular follow-up visits.

Exclusion Criteria:

1. Moderate or severe liver dysfunction (Child-Pugh class B or C);
2. Spontaneous bleeding tendency, such as coagulation disorders or thrombocytopenia (PLT<20×10^9/L);
3. Contraindications to anticoagulant drugs, including allergy to anticoagulants, clinically significant active bleeding, significant risk of major bleeding due to lesions or conditions, significantly abnormal coagulation function, liver disease with clinically relevant bleeding risk, thrombocytopenia, etc., as determined by the attending physician;
4. High-risk pulmonary embolism requiring thrombolysis;
5. Patients currently participating in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Special populations of PTE patients who are elderly, have renal insufficiency, or have concomitant malignancies.
Sampling Method: Probability Sample
Enrollment: 4700 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Major bleeding | From enrollment to 12 months after anticoagulant therapy
  1. Fatal bleeding, and/or
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or
  3. Bleeding causing a fall in hemoglobin level of 20 g L-1 (1.24 mmol L-1) or more, or leading to transfusion of two or more units of whole blood or red cells.
Clinically relevant non-major bleeding | From enrollment to 12 months after anticoagulant therapy
  Any sign or symptom of hemorrhage (e.g., more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for the ISTH definition of major bleeding but does meet at least one of the following criteria:
  i requiring medical intervention by a healthcare professional ii leading to hospitalization or increased level of care iii prompting a face to face (i.e., not just a telephone or electronic communication) evaluation
Recurrent VTE | From enrollment to 12 months after anticoagulant therapy
  Radiologically confirmed recurrent deep vein thrombosis, fatal or non-fatal pulmonary embolism

SECONDARY OUTCOMES:
All-cause mortality | From enrollment to 12 months after anticoagulant therapy
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Pengbo Deng, MD, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China